CLINICAL TRIAL: NCT04253015
Title: A Post-Authorisation Safety Study Patient Registry of Patients With High-risk Neuroblastoma Being Treated With the Monoclonal Antibody Dinutuximab Beta
Brief Title: A Post-Authorisation Safety Study Patient Registry of Patients With Neuroblastoma Being Treated With Dinutuximab Beta
Status: Recruiting | Type: Observational
Sponsor: RECORDATI GROUP (Industry)
Collaborators: United BioSource, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: EUSA DB 0001
Record Dates: First submitted 2020-01-27; First posted 2020-02-05 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Neuroblastoma
Keywords: Tumour; Brain tumour; Paediatrics
MeSH Terms: conditions — Neuroblastoma; Neoplasms; Brain Neoplasms | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Data-collection — Data will be collected on dose, total cumulative amount of dinutuximab beta per course, dose interruptions, dose discontinuations, prophylactic treatment, use of all concomitant analgesia, assessments of pain, and occurrence of neurotoxicity, visual impairment, capillary leak syndrome, cardiovascular events and hypersensitivity reactions and other AEs.

SUMMARY:
This is a non-interventional, multi-national, observational, prospective patient registry to further evaluate the effectiveness and safety of dinutuximab beta - a monoclonal immunoglobulin G 1 (IgG1) antibody, to obtain information on survival, pain severity and incidence of neuro-toxicity, visual impairment, capillary leak syndrome, cardiovascular events, hypersensitivity reactions and long-term safety.

DETAILED DESCRIPTION:
Rationale and Background:

Neuroblastoma, is the most common extra-cranial solid tumour in children. Most patients with neuroblastoma are diagnosed under the age of 5 years and most present with metastatic disease and/or high-risk features. Despite the introduction of novel treatment strategies, including high-dose chemotherapy followed by autologous stem cell transplantation (ASCT), the outcome of these patients remains poor.

Dinutuximab beta is a chimeric monoclonal immunoglobulin G 1 (IgG1) antibody that is specifically directed against the carbohydrate moiety of disialoganglioside antigen (GD2), which is overexpressed on neuroblastoma cells. By binding to neuroblastoma cells, dinutuximab beta can induce both complement dependent cytotoxicity (CDC) and antibody dependent cell-mediated cytotoxicity (ADCC).

The efficacy of dinutuximab beta has been evaluated in a randomised controlled trial comparing the administration of dinutuximab beta with or without interleukin 2 (IL-2) in the first-line treatment of patients with high-risk neuroblastoma and in two singlearm studies in the relapsed/refractory setting. The efficacy and safety of dinutuximab beta will further be evaluated in this registry that will provide information on survival, pain severity and incidence of neurotoxicity, visual impairment, capillary leak syndrome, cardiovascular events, hypersensitivity reactions and long-term safety.

Study Design:

This is a non-interventional, multi-national, observational, prospective patient registry of patients with high-risk neuroblastoma being treated with the monoclonal antibody dinutuximab beta. The efficacy and safety of dinutuximab beta will further be evaluated in this registry that will provide information on survival, pain severity and incidence of neurotoxicity, visual impairment, capillary leak syndrome, cardiovascular events, hypersensitivity reactions and long-term safety.

Research Questions and Objectives:

Primary objectives:

* To assess pain severity and use of analgesics during the period of first dose of dinutuximab beta to end of last 35 day course of the 5th cycle of treatment
* To assess the incidence of neurotoxicity, visual impairment, capillary leak syndrome, cardiovascular events and hypersensitivity reactions
* To assess the long term safety profile

Secondary objectives:

* Progression free survival (PFS) in patients treated with dinutuximab beta.
* Event Free Survival (EFS) in patients treated with dinutuximab beta
* Overall survival (OS) in patients treated with dinutuximab beta

Population:

Patients diagnosed with high-risk neuroblastoma who are starting treatment with dinutuximab beta in the standard clinical practice setting or participating in a clinical trial where dinutuximab beta is provided according to the indication as per the country/regional marketing authorisation, provide consent/assent and are willing to be followed up for up to 10 years.

Study Size:

It is planned to enroll a sufficient number of patients (estimated at 125) such that 100 patients will have completed all five treatment courses of dinutuximab beta. It is anticipated that this will result in 40-50 patients who are progression free at 10 years.

Data Sources:

Data will be collected from physicians using an electronic data capture (EDC) system. The electronic case report forms (eCRFs) will be designed to gather data from the medical records at baseline, during treatment and at normal clinical practice follow up visits.

Data Analysis:

The safety analysis set, containing all patients treated with at least one dose of dinutuximab beta will be considered for safety and efficacy analyses. All baseline, treatment period and follow up characteristics will be summarized using descriptive statistics. Endpoints addressing primary and secondary analysis will include 95% confidence intervals (CIs) including the Clopper Pearson method for binomial, log-log transform for survival. OS, PFS and EFS will be analysed using Kaplan-Meier methods.

Variables:

Baseline (prior to start of treatment): Demographics, clinical trial participation, neuroblastoma disease history, and presence or absence of neurotoxicity, visual impairment, and cardiovascular abnormality.

Treatment period (up to end of last 35 day course of 5th cycle of treatment):

Dosing regimen, total cumulative amount of dinutuximab beta per course, concomitant medications during course (IL-2, retinoic acid and/or antihistamines), daily analgesics (opioids, gabapentin/ pregabalin and/or non-opioid analgesics and other neuropathic pain treatments), daily pain assessment during infusion of dinutuximab beta, occurrence of neurotoxicity, visual impairment, capillary leak syndrome, cardiovascular events, and hypersensitivity reactions, adverse events (AEs)/serious adverse events (SAEs) treatment interruptions and discontinuations, progression of disease, date and cause of death, reason for study withdrawal (if applicable) Follow up (from end of last 35 day course of 5th cycle of treatment): Status of neurotoxicity, visual impairment, cardiovascular events, (resolved, not resolved), SAEs and adverse drug reaction (ADRs), progression of disease, date and cause of death, reason for study withdrawal (if applicable).

ELIGIBILITY:
Inclusion Criteria:

Patients meeting the following criteria will be considered for inclusion into the registry:

* Patients diagnosed with high-risk neuroblastoma and starting treatment with commercially available dinutuximab beta OR
* Patients diagnosed with high-risk neuroblastoma and starting treatment with dinutuximab beta in a clinical trial where dinutuximab beta is provided according to the country/regional marketing authorisation AND
* Appropriate consent/assent has been obtained for participation in the registry with a willingness to be followed up for up to 10 years.

Exclusion Criteria:

Patient will not be eligible for inclusion if the following criterion applies:

* Patients commencing dinutuximab beta within a clinical trial where the product is being provided outside of the country/regional marketing authorisation OR
* Appropriate consent/assent has not been obtained for participation in the registry or patient/legal representative is not willing for the patient be followed up for up to 10 years.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients diagnosed with high-risk neuroblastoma who are starting treatment with dinutuximab beta in the standard clinical practice setting or participating in a clinical trial where dinutuximab beta is provided according to the indication as per the country/regional marketing authorisation, provide consent/assent and are willing to be followed up for up to 10 years. Centers who treat neuroblastoma patients with dinutuximab beta will be invited to participate in the registry. This includes networks such as the Society of Paediatric Oncology for the Treatment of Neuroblastoma (SIOPEN) in Europe.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2019-09-30 (Actual); Primary Completion 2032-03-31 (Estimated); Study Completion 2032-06-15 (Estimated)

PRIMARY OUTCOMES:
Assessment of the severity of pain experienced by participants during treatment with dinutuximab beta | First dose of dinutuximab beta to the end of the last 35 day course of the 5th cycle of treatment (each cycle is 35 days)
  Assessment of pain severity experienced by participants during the period of first dose of dinutuximab beta to the end of last 35 day course of 5th cycle of treatment
Number of participants using analgesics during treatment with dinutuximab beta | First dose of dinutuximab beta to the end of the last 35 day course of the 5th cycle of treatment (each cycle is 35 days)
  Use of analgesics during the period of first dose of dinutuximab beta to end of last 35 day course of 5th cycle of treatment
Incidence of neurotoxicity, visual impairment, capillary leak syndrome, cardiovascular events and hypersensitivity reactions | First dose of dinutuximab beta to the end of the last 35 day course of the 5th cycle of treatment (each cycle is 35 days)
  Incidence of neurotoxicity, visual impairment, capillary leak syndrome, cardiovascular events and hypersensitivity reactions up to the end of the last 35 day course of 5th cycle of treatment
Number of participants experiencing serious adverse events (SAEs) and adverse drug reactions (ADRs) during treatment with dinutuximab beta | First dose of dinutuximab beta to the end of the last 35 day course of the 5th cycle of treatment (each cycle is 35 days)
  Number of participants experiencing serious adverse events (SAEs) and adverse drug reactions (ADRs) following the end of the last 35 day course of 5th cycle of treatment

SECONDARY OUTCOMES:
Overall Survival (OS) | First dose of dinutuximab beta to the end of the last 35 day course of the 5th cycle of treatment (each cycle is 35 days)
  Overall Survival (OS) following the end of the last 35 day course of 5th cycle of treatment
Progression free survival (PFS) | First dose of dinutuximab beta to the end of the last 35 day course of the 5th cycle of treatment (each cycle is 35 days)
  Progression free survival (PFS) following the end of the last 35 day course of 5th cycle of treatment
Event Free Survival (EFS) | First dose of dinutuximab beta to the end of the last 35 day course of the 5th cycle of treatment (each cycle is 35 days)
  Event Free Survival (EFS) following the end of the last 35 day course of 5th cycle of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jose-Luis Garcia, Study Director — EUSA Pharma (UK) Limited
Locations (13):
- St. Anna Kinderkrebsforschung, Vienna, Vienna, Austria
- France (4):
  - Centre Oscar Lambret, Lille
  - Hôpital de la Timone, Hôpital des Enfants, Marseille
  - Institut Curie, Paris
  - Institut Gustave Roussy, Villejuif
- Germany (2):
  - Charité Berlin, Berlin
  - Universitätsmedizin Greifswald, Greifswald
- IRCCS Istituto Giannina Gaslini, Genova, Italy
- Uniwersytecki Szpital Dziecięcy, Krakow, Poland
- Hospital Universitario y Politecnico La Fe Avenida Fernando Abril Martorell, Valencia, Spain
- United Kingdom (3):
  - The Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne, Newcastle
  - Birmingham Children's Hospital, Birmingham
  - University Hospital Southampton, Southampton

IPD SHARING:
Plan to Share IPD: No